CLINICAL TRIAL: NCT07152106
Title: The Impact of Amniotic Fluid on the Development and Microbial Colonization of the Preterm Intestinal Tract: the AMFIBIE Study
Brief Title: Amniotic Fluid & the Preterm Gut
Acronym: AMFIBIE
Status: Recruiting | Type: Observational
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Hendrik Niemarkt, Principal Investigator, Maxima Medical Center
Other Study IDs: NL86579.018.24; NL86579.018.24 (Other: CCMO)
Record Dates: First submitted 2025-08-20; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Chorioamnionitis; Chorioamnionitis Affecting Fetus or Newborn; Necrotizing Enterocolitis of Newborn; Neonatal Sepsis, Early-Onset; Neonatal Sepsis, Late-Onset; Fetal Growth Restriction (FGR); Preterm Birth Complication; Prematurity Complications
MeSH Terms: conditions — Chorioamnionitis; Neonatal Sepsis; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Amniotic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Total cohort consists of: 1) study group - gestational age 24+0/7-27+6/7 weeks, 2) reference/control group: <24+0/7 weeks and 28+0/7-40+6/7 weeks

SUMMARY:
Background:

Necrotizing enterocolitis (NEC) and sepsis in preterm infants have been linked to intestinal immaturity and preclinical gut microbiota alterations. An important yet understudied contributor in the development of the gastrointestinal tract (GIT) is amniotic fluid (AF). Knowledge is lacking on the critical shifts that may occur in AF in extremely preterm birth. The aim of the current study is to assess the composition of AF using advanced biomedical techniques. Secondary objectives are to assess AF profiles of infants with chorioamnionitis (CAM) and/or fetal growth restriction (FGR), assess key metabolites across gestation, correlate AF profiles with neonatal outcomes, and explore associations with early gut microbiota.

Methods:

ln this multicenter, prospective, cohort study, AF (~5 mL) will be collected from obstetric patients delivering their infants extremely preterm (gestational age (GA) 24+0/7-27+6/7 weeks, n=125), either during vaginal delivery or cesarean section (CS). Additionally, AF samples will be collected from a reference group (n=150), including early midtrimester (GA <23+/7 weeks), very early and moderate to late preterm (GA 28+0/6-36+6/7 weeks), and full-term pregnancies (GA 37+0/7-41+6/7 weeks). Thorough characterization of AF will be conducted, including microbial profiling and metabolomics. Microbiota profiling of neonatal fecal samples will be conducted to assess the association between AF and early neonatal gut colonization patterns.

Discussion and expected results:

AF profiles associated with CAM and/or FGR in extremely preterm infants are expected to be identified, as well as relevant associations with neonatal health outcomes (including NEC and sepsis) and early neonatal gut colonization patterns. The current study will not only increase the understanding of the GIT development and the pathogenesis of NEC and sepsis but may also aid in the identification of high-risk infants. In the future, these findings may facilitate early targeted microbiota-based interventions to prevent disease progression and ultimately improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥16 years
* Written informed consent
* Successful collection of amniotic fluid

Exclusion Criteria:

* Pregnancies complicated by fetal congenital and/or chromosomal abnormalities.
* Insufficient proficiency of Dutch or English language

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants included in the study group must be born between 24+0/7 and 27+6/7 weeks. AF samples are also collected from a reference group, including early midtrimester (GA ≤23+6/7 weeks), very and moderate to late preterm (GA 28+0/7-36+6/7 weeks), and full-term pregnancies (GA 37+0/7-41+6/7 weeks).
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
AF & preterm birth | Baseline
  Microbial & metabolic composition of amniotic fluid in extremely preterm birth

SECONDARY OUTCOMES:
AF profiles & chorioamnionitis | Baseline
  Characterizion of AF profiles in infants exposed to chorioamnionitis
AF & fetal growth restriction | Baseline
  Characterizion of AF profiles in infants with fetal growth restriction
AF & neonatal gut microbiota | For AF baseline measurement, for neonatal gut microbiota composition at t=0, t=7, t=14, t=21, and t=28 (postnatal days)
  To correlate composition of amniotic fluid to neonatal gut microbiota in first month of life

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Máxima Medical Center, Veldhoven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Puri K, Taft DH, Ambalavanan N, Schibler KR, Morrow AL, Kallapur SG. Association of Chorioamnionitis with Aberrant Neonatal Gut Colonization and Adverse Clinical Outcomes. PLoS One. 2016 Sep 22;11(9):e0162734. doi: 10.1371/journal.pone.0162734. eCollection 2016. PMID 27658190
- [Result] de Kroon RR, de Baat T, Senger S, van Weissenbruch MM. Amniotic Fluid: A Perspective on Promising Advances in the Prevention and Treatment of Necrotizing Enterocolitis. Front Pediatr. 2022 Mar 14;10:859805. doi: 10.3389/fped.2022.859805. eCollection 2022. PMID 35359891
- [Result] Dasgupta S, Arya S, Choudhary S, Jain SK. Amniotic fluid: Source of trophic factors for the developing intestine. World J Gastrointest Pathophysiol. 2016 Feb 15;7(1):38-47. doi: 10.4291/wjgp.v7.i1.38. PMID 26909227
- [Derived] de Kroon RR, van Weelden S, Monen L, Bakker P, Pajkrt E, Struys EA, Budding AE, de Meij T, Niemarkt HJ, van Weissenbruch MM. The impact of AMniotic FluId on the development and microBIal colonization of the prEterm intestinal tract (AMFIBIE): study protocol for a multicenter prospective cohort study. Front Pediatr. 2026 Jan 12;13:1721519. doi: 10.3389/fped.2025.1721519. eCollection 2025. PMID 41602874

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT07152106/Prot_SAP_000.pdf